CLINICAL TRIAL: NCT06906237
Title: Scarless Advanced Breast Extended Oncoplasty: The ScarABEO Study
Acronym: ScarABEO
Status: Recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: CET ANV 2024-23
Record Dates: First submitted 2025-03-07; First posted 2025-04-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Oncoplastic Breast Surgery; Oncoplastic Breast-conserving Surgery; Chest Wall Perforator Flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast conserving surgery followed by radiotherapy is the gold standard treatment for early breast cancer. Cases with unfavorable tumor volume to breast volume ratio or challenging localizations are at higher risk of margin infiltration or poor aesthetic outcomes. While margin infiltration represents one of the strongest predictors of local recurrence, unappealing cosmetic results may significantly impair survivors' quality of life. Over the past two decades, the adoption of oncoplastic breast conserving surgery (OBCS) techniques has shown promise in improving both oncological and aesthetic outcomes after breast cancer surgery. Partial breast volume reconstruction (PBR) after OBCS is obtained through volume displacement (which involves remodelling and redistributing glandular tissue) and volume replacement (when the volume used to reconstruct the defect comes from an extramammary site) techniques.

One of the greatest examples of volume replacement techniques in breast surgery involves the use of chest wall perforator flaps (CWPF). The use of these well-vascularized dermo-adipose flaps offers oncologically safe wide resection while obtaining excellent cosmetic outcomes. It is particularly suitable for patients with non-ptotic small to medium-sized breasts and cases with an unfavorable tumor volume to breast volume ratio. CWPFs can decrease mastectomy rates in breast cancer surgery, thus avoiding the disadvantages associated with implant-based reconstruction. Consequently, the need of contralateral simmetrization is also diminished.

CWPFs are vascularized by perforator arteries that arise from the chest wall (mainly branches of the axillary artery, or intercostal arteries deriving from the internal mammary artery). While cadaver labs and radiologic studies demonstrated a reliable and coherent localization of perforator arteries, the use of Doppler Ultrasound is often required to localize the perforators and test their reliability. Compared to the traditional myocutaneous flaps (such as the latissimus dorsi flap), CWPFs spare the underlying muscles minimizing donor site morbidity and enabling rapid post-operative recovery, low post-operative complication rates, post-operative pain, and loss of function. All these advantages may result in high levels of patients' satisfaction. Additionally, CWPFs avoid the microsurgical anastomoses required for free flaps.

All breast quadrants defects could be restored with CWPFs, with the Thoraco-Dorsal Artery Perforator (TDAP), Lateral-Thoracic Artery Perforators (LTAP) and Lateral Intercostal Artery Perforator (LICAP) Flaps particularly suitable for reconstructing lateral quadrant; the Anterior Intercostal Artery Perforator (AICAP) Flap for the lower quadrants and the Internal Mammary Artery Perforator (IMAP) Flaps for volume defects at inner quadrants.

Although existing literature reports promising results, the use of CWPFs remains emerging, and OBCS with CWPFs is currently limited to select high-volume breast centers. The collection of robust clinical data is essential to validate these potential advantages and facilitate the broader adoption of this technique.

This multicentric retrospective observational study aims to collect evidence about the surgical and oncological outcomes of OBCS with CWPFs, to evaluate the potential benefits associated with the use of this innovative technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with BCS combined with CWPFs for primary stage I-III invasive cancer (IC) or ductal carcinoma in situ (DCIS);
* Patients treated during the last 10 years (2015-2025);
* Patients aged 18 years or more;
* Cases with at least one-year follow-up.

Exclusion Criteria:

* Male Patients;
* Patients aged less than 18 years;
* Patients who underwent traditional breast conserving surgery or OBCS with displacement techniques;
* Patients who underwent mastectomy;
* Patients who underwent implant-based reconstruction;
* Patients with unresectable breast cancer or metastatic disease;
* Patients who were lost during follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female Patients who underwent OBCS with CWPFs for breast cancer, with at least one-year follow-up
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Margin infiltration rate | Perioperative
  Margin infiltration rate in Patients with breast cancer or ductal carcinoma in situ who underwent Oncoplastic Breast Conserving Surgery with Chest Perforator Flaps

SECONDARY OUTCOMES:
Re-excisions rate | Up to 24 weeks
  Re-excisions rate due to positive margins rate on surgical specimen
Total resection volume and final breast volume ratio | Perioperative
Post-operative complication rates | Up to 24 weeks
Post-operative breast symmetry | One year
Disease-free survival | Two years
Overall Survival | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Veneto Institute of Oncology, Padua, Italy

IPD SHARING:
Plan to Share IPD: No